CLINICAL TRIAL: NCT02800213
Title: Single Rescuer Ventilation Using a Bag Valve Mask With Supplemental External Handle Versus Standard Bag Valve Mask in a Manikin Model: A Randomized Crossover Trial
Brief Title: Ventilation Using a Bag Valve Mask With Supplemental External Handle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael D. April, Assistant Director for Research, Emergency Medicine Residency, Brooke Army Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C.2016.136e
Record Dates: First submitted 2016-06-12; First posted 2016-06-15 (Estimated); Results first posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Apnea
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified Ambu Spur II bag mask first (Experimental): A health volunteer uses a modified Ambu Spur II bag valve mask with integrated internal handle (experimental device, not yet FDA approved) to deliver 10 breaths per minute for 3 minutes to a manikin (IngMar RespiTrainer manikin model). Volunteer then repeats the procedures using a conventional Ambu Spur II bag valve mask.
  Interventions: Device: Modified Ambu Spur II bag valve mask; Device: Conventional Ambu Spur II bag valve mask
- Conventional Ambu Spur II bag mask first (Active Comparator): A health volunteer uses a conventional Ambu Spur II bag valve mask to deliver 10 breaths per minute for 3 minutes to a manikin (IngMar RespiTrainer manikin model). Volunteer then repeats the procedures using a modified Ambu Spur II bag valve mask.
  Interventions: Device: Modified Ambu Spur II bag valve mask; Device: Conventional Ambu Spur II bag valve mask

INTERVENTIONS:
Device: Modified Ambu Spur II bag valve mask — Subjects deliver breaths to manikin (IngMar RespiTrainer manikin model) a modified Ambu Spur II bag valve mask with a supplemental external handle
Device: Conventional Ambu Spur II bag valve mask — Subjects deliver breaths to manikin (IngMar RespiTrainer manikin model) a conventional Ambu Spur II bag valve mask

SUMMARY:
Investigators compared tidal volumes for single rescuer ventilation using a modified bag valve mask with a supplemental external handle versus a conventional bag valve mask in a manikin model.

DETAILED DESCRIPTION:
This was a prospective, randomized, crossover study to assess the tidal volume delivered using a standard and modified bag valve mask (BVM) device in a manikin airway model. The modified device comprised a standard bag valve mask with supplemental external bar. Data was collected during May 2016 at the San Antonio Military Medical Center. Emergency medicine providers (physicians, physician assistants, residents, nurses, medics) were randomized to device order. Prior to participation each participant filled out a survey indicating their job status, gender, years of medical experience, and experience level with BVM ventilation. Hand grip strength and size (length, width, span) were measured. Each participant was then asked to provide BVM ventilation using the assigned devices at a rate of 10 breaths per minute for 3 minutes for a total of 30 breaths. Tidal volume of each delivered breath was recorded in milliliters. After a 3 minute rest period, testing was repeated with the second device. After ventilation with each device, participants completed an anonymous questionnaire that used a Likert scale to assess perceived qualities of the modified device including ease of use, ability to provide a superior mask seal, willingness to use in an emergency situation, and overall preference between the two devices. Each participant served as his/her own control.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Department healthy volunteers (physician assistants, residents, paramedics, nurses, medics, respiratory therapists).

Exclusion Criteria:

* Not trained in basic life support

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D April, MD, DPhil, Study Director — Brooke Army Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davidovic L, LaCovey D, Pitetti RD. Comparison of 1- versus 2-person bag-valve-mask techniques for manikin ventilation of infants and children. Ann Emerg Med. 2005 Jul;46(1):37-42. doi: 10.1016/j.annemergmed.2005.02.005. PMID 15988424
- [Background] Braude DA, Tawil I, Gerstein NS, Carey MC, Petersen TR. Comparison of bag-valve-mask hand-sealing techniques in a simulated model. Ann Emerg Med. 2014 Jun;63(6):784-5. doi: 10.1016/j.annemergmed.2014.01.037. No abstract available. PMID 24841402
- [Background] Otten D, Liao MM, Wolken R, Douglas IS, Mishra R, Kao A, Barrett W, Drasler E, Byyny RL, Haukoos JS. Comparison of bag-valve-mask hand-sealing techniques in a simulated model. Ann Emerg Med. 2014 Jan;63(1):6-12.e3. doi: 10.1016/j.annemergmed.2013.07.014. Epub 2013 Aug 9. PMID 23937957
- [Background] Amack AJ, Barber GA, Ng PC, Smith TB, April MD. Comparison of Ventilation With One-Handed Mask Seal With an Intraoral Mask Versus Conventional Cuffed Face Mask in a Cadaver Model: A Randomized Crossover Trial. Ann Emerg Med. 2017 Jan;69(1):12-17. doi: 10.1016/j.annemergmed.2016.04.017. Epub 2016 May 27. PMID 27238825

RESULTS

PARTICIPANT FLOW:
Groups:
- Modified Then Conventional Ambu Spur II Bag Valve Mask: A health volunteer uses a modified Ambu Spur II bag valve mask with integrated internal handle (experimental device, not yet FDA approved) to deliver 10 breaths per minute for 3 minutes to a manikin (IngMar RespiTrainer manikin model).
  Modified Ambu Spur II bag valve mask: Subjects deliver breaths to manikin (IngMar RespiTrainer manikin model) a modified Ambu Spur II bag valve mask with a supplemental external handle.
  After completion, subjects repeat all these procedures using a conventional Ambu Spur II bag valve mask.
- Conventional Then Modified Ambu Spur II Bag Valve Mask: A health volunteer uses a conventional Ambu Spur II bag valve mask to deliver 10 breaths per minute for 3 minutes to a manikin (IngMar RespiTrainer manikin model).
  Conventional Ambu Spur II bag valve mask: Subjects deliver breaths to manikin (IngMar RespiTrainer manikin model) a conventional Ambu Spur II bag valve mask
  After completion, subjects repeat all these procedures using the modified Ambu Spur II bag valve mask.
Period: First Intervention
Arm/Group | Modified Then Conventional Ambu Spur II Bag Valve Mask | Conventional Then Modified Ambu Spur II Bag Valve Mask
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Modified Then Conventional Ambu Spur II Bag Valve Mask | Conventional Then Modified Ambu Spur II Bag Valve Mask
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Conventional Then Modified Ambu Spur II Bag Valve Mask: A health volunteer uses a conventional Ambu Spur II bag valve mask to deliver 10 breaths per minute for 3 minutes to a manikin (IngMar RespiTrainer manikin model).
  Conventional Ambu Spur II bag valve mask: Subjects deliver breaths to manikin (IngMar RespiTrainer manikin model) a conventional Ambu Spur II bag valve mask.
  After completion, subjects repeat all these procedures using the modified Ambu Spur II bag valve mask.
- Total: Total of all reporting groups
Arm/Group | Modified Then Conventional Ambu Spur II Bag Valve Mask | Conventional Then Modified Ambu Spur II Bag Valve Mask | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 35 | 70
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 19 | 19 | 38
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Received Tidal Volume
Description: Mean received tidal volume for 30 breaths delivered by the subjects over three minutes as measured via the RespiTrainer Advance manikin model monitor output.
Time Frame: 3 minutes
Measure: Mean (95% Confidence Interval); unit: milliliters
Groups:
- Modified Ambu Spur II Bag Valve Mask: A health volunteer uses a modified Ambu Spur II bag valve mask with integrated internal handle (experimental device, not yet FDA approved) to deliver 10 breaths per minute for 3 minutes to a manikin (IngMar RespiTrainer manikin model).
  Modified Ambu Spur II bag valve mask: Subjects deliver breaths to manikin (IngMar RespiTrainer manikin model) a modified Ambu Spur II bag valve mask with a supplemental external handle.
  After completion, subjects repeat all these procedures using a conventional Ambu Spur II bag valve mask.
- Conventional Bag Valve Mask: A health volunteer uses a conventional Ambu Spur II bag valve mask to deliver 10 breaths per minute for 3 minutes to a manikin (IngMar RespiTrainer manikin model).
  Conventional Ambu Spur II bag valve mask: Subjects deliver breaths to manikin (IngMar RespiTrainer manikin model) a conventional Ambu Spur II bag valve mask.
  After completion, subjects repeat all these procedures using the modified Ambu Spur II bag valve mask.
Arm/Group | Modified Ambu Spur II Bag Valve Mask | Conventional Bag Valve Mask
Number analyzed (Participants) | 70 | 70
milliliters | 662 [611 to 707] | 681 [635 to 731]
Statistical Analysis 1: Comparison: Modified Ambu Spur II Bag Valve Mask vs Conventional Bag Valve Mask; Test type: Superiority; p = 0.280, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 hour
Groups:
- Conventional Ambu Spur II Bag Valve Mask: A health volunteer uses a conventional Ambu Spur II bag valve mask to deliver 10 breaths per minute for 3 minutes to a manikin (IngMar RespiTrainer manikin model).
  Conventional Ambu Spur II bag valve mask: Subjects deliver breaths to manikin (IngMar RespiTrainer manikin model) a conventional Ambu Spur II bag valve mask.
  After completion, subjects repeat all these procedures using the modified Ambu Spur II bag valve mask.
Arm/Group | Modified Ambu Spur II Bag Valve Mask | Conventional Ambu Spur II Bag Valve Mask
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No